CLINICAL TRIAL: NCT02868814
Title: The Efficacy and Safety of Pregabalin Release Tablets for the Treatment of Fibromyalgia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-PRBL-FM
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 330mg/day (Experimental): 330 mg QD taken orally,1 pills once ,one time a day in an hour after meals, oral administration for 15 weeks (3 week titration and 12-week fixed dose)
  Interventions: Drug: Pregabalin Release Tablets
- 495mg/day (Experimental): 495 mg QD taken orally,2 pills once ,one time a day in an hour after meals, oral administration for 15 weeks (3 week titration and 12-week fixed dose)
  Interventions: Drug: Pregabalin Release Tablets
- Placebo (Placebo Comparator): 1 or 2 pills once ,one time a day in an hour after meals, oral administration for 15 weeks (3 week titration and 12-week fixed dose)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin Release Tablets
  Arms: 330mg/day
Drug: Pregabalin Release Tablets
  Arms: 495mg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Efficacy and safety of pregabalin sustained release tablets versus placebo for fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the 1990 American College of Rheumatology (ACR) criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites).

Patients who completed at least 4 pain diaries within the last 7 days and the average pain score must have been ≥4, and had a score of ≥40 mm on the Visual Analogue Scale (VAS) at screening and randomization .

Exclusion Criteria:

* Patients with other severe pain that may confound assessment or self-evaluation of the pain associated with fibromyalgia.

Patients with any inflammatory muscle or rheumatologic disease other than fibromyalgia, active infections, or untreated endocrine disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean pain score diary at Endpoint | Baseline and 15 weeks
  derived from the subject's daily pain

SECONDARY OUTCOMES:
Change from baseline in FIQ scores at Weeks 15 | Baseline and Weeks 15
Change from baseline in SF-36 scores at Weeks 15 | Baseline and Weeks 15
Change from baseline in HADS scores at Weeks 15 | Baseline and Weeks 15
Change from baseline in MOS-SS scores at Weeks 15 | Baseline and Weeks 15
Quality of Sleep Score from the Daily Sleep Diary | up to 15 weeks
Mean pain score from the subject's daily pain | up to 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xiehe Hospital of Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided